CLINICAL TRIAL: NCT03075579
Title: Atomoxetine, Diurnal Profiles of Cortisol and α-amylase, Possible Biological Markers of Treatment Success
Brief Title: Atomoxetine, Diurnal Profiles of Cortisol and α-amylase
Acronym: ADHDstress
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Praxis für kleine und grosse Leute (Other)
Collaborators: Dr med Kurt von Siebenthal, Facharztpraxis für Pädiatrie, Winterthur, Switzerland (Unknown); Dr med Roland Kägi, Facharztpraxis für Pädiatrie, Zurich, Switzerland (Unknown); Dr med Corrado Garbazza, University of Basle, Switzerland (Unknown); Prof Vivette Glover, Imperial College London, UK (Unknown); Prof Alina Rodriguez, University of Lincoln, UK (Unknown)
Responsible Party: Principal Investigator, Martin Kammerer MD PhD, Principal Investigator, Praxis für kleine und grosse Leute
Other Study IDs: ADHDstress
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: ADHD
Keywords: ADHD, cortisol, α-amylase, actometer
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Drug: Medication Other — medication of atomoxetine
  Other Names: atomoxetine
Device: motor measurement and saliva collection — motor measurement by actometer and saliva collection for measurement of saliva cortisol and saliva alpha amylase

SUMMARY:
Diurnal profiles of markers of the stress system are increasingly recognized as biomarkers of different kinds of depression and related states. They may also serve as markers of treatment success. However, this has not yet been studied in attention deficit disorder (ADHD). Especially, there is a paucity of research into the effect of ADHD medication on the diurnal profiles of cortisol as marker of the hypothalamic pituitary adrenal (HPA) system and of amylase as marker of the sympathetic adrenomedullar (SAM) system.

The investigators propose a within subjects design with probands of a narrow age range (seven to ten years of age, same sex: boys only) in order to get first information about whether there is an effect of atomoxetine on these diurnal profiles of cortisol and amylase, what kind of effect it is and whether this effect is related to treatment success. The investigators control for motor activity by using actometer measurements.

DETAILED DESCRIPTION:
Scientific and clinical Background

There is very good evidence that the hypothalamic-pituitary- adrenal (HPA) axis is disturbed in depression. There is some evidence that the stress system also plays a role in attention deficit disorder (ADHD ) (O'Connor, Heron et al. 2002).

The investigators have shown that motor activity and attention deficit/concentration are core symptoms of depression (Kammerer, Marks et al. 2009; Kammerer 2010). These symptoms are also the core symptoms of attention deficit hyperkinetic disorder (ADHD). There is increasing evidence that the diurnal variation of markers of the stress system (e.g. salivary cortisol for the hypothalamic pituitary adrenal (HPA) axis, salivary amylase for the sympathetic adrenomedullar (SAM) axis) reveal characteristics of different types of depression, e.g. atypical depression (Tops, Riese et al. 2008), post partum depression (Tops, Riese et al. 2008; Taylor, Glover et al. 2009) and related states, e.g. posttraumatic stress disorder (PTSD) (Wessa, Rohleder et al. 2006) and chronic fatigue syndrome (Roberts, Wessely et al. 2004).

There is some evidence that the saliva cortisol levels and the cortisol awakening rise may be markers of treatment success (Roberts, Papadopoulos et al. 2009). Salivary cortisol and salivary amylase are easy to study as only saliva is needed. (Clow, Hucklebridge et al.; Kirschbaum and Hellhammer 1989; O'Donnell, Kammerer et al. 2009). The investigators have tested saliva amylase, found it to be robust and a useful marker for the function of the SAM system (O'Donnell, Kammerer et al. 2009).

However there is still insufficient research into the diurnal profile of cortisol and amylase with children suffering from ADHD. This causes a serious lack of information for both clinical child and adolescent psychiatry and paediatrics as well as for the research community.

Atomoxetine was originally developed to be used as an antidepressant and shows an excellent therapeutic effect on attention deficit and hyperactivity with children suffering from ADHD. It is a selective re-uptake inhibitor of noradrenaline from the synaptic cavity (NARI).

Research into the possible effect of medication with Atomoxetine in children on their diurnal profile of cortisol and amylase has - to the investigators' best knowledge - not been carried out. The possible effect on the diurnal profile of cortisol and amylase could be linked to treatment success in general and to improvement of individual symptoms of ADHD. It may also contribute to a better understanding of possible side effects.

The investigators propose a study - with a within subjects design - with five times daily saliva collection on two consecutive weekdays before medication commences. Measurements will be repeated in weeks one, four and twelve of medication of Atomoxetine. Additional questionnaire data collection (Conners, CBCL) and, if feasible, testing (KI TAP) will be carried out.

The study will provide insight into possible effects of the compound (Atomoxetine) on the stress system. It may identify easily measurable biological markers of treatment success, and provide research into possible markers of respondents and non respondents. The investigators control for motor activity by using actometers.

Hypotheses to be tested

1. The cortisol awakening reaction (CAR) will be significantly different before, immediately after and four and twelve weeks after begin of the mediation of Atomoxetine with boys aged seven to ten.
2. The overall cortisol level will be different at the three measurement time points from each other.
3. The diurnal profile of salivary amylase and the overall amylase level will be significantly different from each other at the three measurement time points.
4. There will be a group effect regarding the diurnal profile distinguishing responders to Atomoxetine (response=50%reduction of symptoms) from non responders.

Plan of Research

Ethical approval

The protocol has obtained approval by the relevant ethical committees prior to begin of the study.

Location

A network of paediatrician's n Switzerland.

Subjects and tests

Eligibility criteria:

Boys are eligible, age seven to ten, without comorbid psychiatric and/or somatic condition for whom the responsible paediatrician and/or child psychiatrist gives the indication for treatment with Atomoxetine and parents follow this advice. In order to exclude effects of prior psycho pharmacotherapy psychotropic drug naive boys only will be chosen. The diurnal variation seems to change as children grow older (unpublished observations of our group). Therefore, we want to try to get a sample that is as homogenous as possible.

Exclusion criteria:

Suicidal risk, depression, history of epileptic seizures, co morbid psychiatric or somatic conditions, history of psychotropic medication.

Power:

With an n=50 the investigators expect a power of 80% at 5 % significance and an SD of 0.6. In our study of postpartum depression (Taylor et al, 2009) we reached significant differences between the groups with an n= 30 and an n=21.

Sample:

• 50 boys, seven to ten yours of age, with clinical diagnosis of ADHD (ICD 10 or DSMV)

Measurements

Biological measures

Method for measurement of saliva cortisol and saliva amylase:

The same methodology will be applied as in (O'Donnell, Kammerer et al. 2009; Taylor, Glover et al. 2009) Actometer measurements using actometers provided by www.resmed.ch

Psychological measures

Assessment tools for quantifying ADHD symptoms will include the German version of the CPRS-R:L (Conners 1998; Conners, Sitarenios et al. 1998; Conners, Sitarenios et al. 1998), the CTRS-R:L (Conners, Sitarenios et al. 1998), the SDQ, parent and teacher version (Goodman 1997), Achenbach, T.M., & Rescorla, L. A. (2001). Manual for the ASEBA School-Age Forms and Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, and Families. ISBN 0-938565-73-7

ELIGIBILITY:
Inclusion Criteria:

Boys are eligible, age seven to ten, without comorbid psychiatric and/or somatic condition for whom the responsible paediatrician and/or child psychiatrist gives the indication for treatment with atomoxetine.

Exclusion Criteria:

Suicidal risk, depression, history of epileptic seizures, comorbid psychiatric or somatic conditions, history of psychotropic medication.

Ages: 7 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Boys only
Study Population: Boys are eligible, age seven to ten, dignosed with ADHD, without comorbid psychiatric and/or somatic condition for whom the responsible paediatrician and/or child psychiatrist gives the indication for treatment with atomoxetine and the parents accept their advice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
saliva cortisol | 13 weeks
  diurnal profile of saliva cortisol and saliva alpha amylase

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kammerer, MD PHD, Principal Investigator — Praxis fuer kleine und grosse Leute, Rueschlikon, Switzerland and Imperial College London
Locations (2):
- Switzerland (2):
  - Dr med Kurt von Siebenthal, Winterthur, Canton of Zurich
  - Dr med Roland Kägi, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wessa M, Rohleder N, Kirschbaum C, Flor H. Altered cortisol awakening response in posttraumatic stress disorder. Psychoneuroendocrinology. 2006 Feb;31(2):209-15. doi: 10.1016/j.psyneuen.2005.06.010. Epub 2005 Sep 9. PMID 16154709
- [Background] Taylor A, Glover V, Marks M, Kammerer M. Diurnal pattern of cortisol output in postnatal depression. Psychoneuroendocrinology. 2009 Sep;34(8):1184-8. doi: 10.1016/j.psyneuen.2009.03.004. Epub 2009 Apr 29. PMID 19406580
- [Background] O'Donnell K, Kammerer M, O'Reilly R, Taylor A, Glover V. Salivary alpha-amylase stability, diurnal profile and lack of response to the cold hand test in young women. Stress. 2009 Nov;12(6):549-54. doi: 10.3109/10253890902822664. PMID 19658030
- [Background] Roberts AD, Wessely S, Chalder T, Papadopoulos A, Cleare AJ. Salivary cortisol response to awakening in chronic fatigue syndrome. Br J Psychiatry. 2004 Feb;184:136-41. doi: 10.1192/bjp.184.2.136. PMID 14754825
- [Background] Conners CK. Rating scales in attention-deficit/hyperactivity disorder: use in assessment and treatment monitoring. J Clin Psychiatry. 1998;59 Suppl 7:24-30. PMID 9680050
- [Background] Garbazza C, Bromundt V, Eckert A, Brunner DP, Meier F, Hackethal S, Cajochen C. Non-24-Hour Sleep-Wake Disorder Revisited - A Case Study. Front Neurol. 2016 Feb 29;7:17. doi: 10.3389/fneur.2016.00017. eCollection 2016. PMID 26973592
- [Background] Roberts AD, Papadopoulos AS, Wessely S, Chalder T, Cleare AJ. Salivary cortisol output before and after cognitive behavioural therapy for chronic fatigue syndrome. J Affect Disord. 2009 May;115(1-2):280-6. doi: 10.1016/j.jad.2008.09.013. Epub 2008 Oct 19. PMID 18937978
- [Background] O'Connor TG, Heron J, Golding J, Beveridge M, Glover V. Maternal antenatal anxiety and children's behavioural/emotional problems at 4 years. Report from the Avon Longitudinal Study of Parents and Children. Br J Psychiatry. 2002 Jun;180:502-8. doi: 10.1192/bjp.180.6.502. PMID 12042228
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychobiological research: an overview. Neuropsychobiology. 1989;22(3):150-69. doi: 10.1159/000118611. PMID 2485862
- [Background] Kammerer M, Marks MN, Pinard C, Taylor A, von Castelberg B, Kunzli H, Glover V. Symptoms associated with the DSM IV diagnosis of depression in pregnancy and post partum. Arch Womens Ment Health. 2009 Jun;12(3):135-41. doi: 10.1007/s00737-009-0062-9. Epub 2009 Apr 1. PMID 19337702
- [Background] Kammerer M, Glover V, Pinard Anderman C, Kunzli H, Taylor A, von Castelberg B, Marks M. The DSM IV diagnoses of melancholic and atypical depression in pregnancy. Arch Womens Ment Health. 2011 Feb;14(1):43-8. doi: 10.1007/s00737-010-0187-x. Epub 2010 Oct 15. PMID 20949294